CLINICAL TRIAL: NCT06827509
Title: Blood Flow Evaluation After Carotid Surgical Treatment: Carotid Endarterectomy With Patch Repair Versus Eversion Technique
Brief Title: Blood Flow Evaluation After Carotid Surgical Treatment
Acronym: BEAT
Status: Not yet recruiting | Type: Observational
Sponsor: Rijnstate Hospital (Other)
Collaborators: Elisabeth-TweeSteden Ziekenhuis (Other); Medisch Spectrum Twente (Other); Radboud University Medical Center (Other); University of Twente (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-2578
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Carotid Endarterectomy
Keywords: Ultrafast ultrasound flow imaging; Velocity vector imaging; Carotid endarterectomy; Patch repair; Eversion technique

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CEA with patch repair (CEAP): Patients with a carotid artery stenosis that underwent recent conventional carotid endarterectomy with patch repair. Ultrasound measurements were performed 6-8 weeks after CEAP.
  Interventions: Diagnostic Test: Ultrasound-based flow imaging
- CEA with eversion technique (ET): Patients with a carotid artery stenosis that underwent recent carotid endarterectomy with the eversion technique. Ultrasound measurements were performed 6-8 weeks after CEAP.
  Interventions: Diagnostic Test: Ultrasound-based flow imaging

INTERVENTIONS:
Diagnostic Test: Ultrasound-based flow imaging — Ultrasound-based flow imaging (based on blood speckle tracking) of the carotid artery will be acquired at 6-8 weeks after surgery.
  Other Names: Velocity vector imaging; Ultrafast flow imaging

SUMMARY:
Approximately 20% of strokes originate from the rupture of an atherosclerotic plaque in the carotid artery. Surgical revascularization, i.e. carotid endarterectomy (CEA), is the treatment of choice for patients with a symptomatic carotid stenosis each year about 3,000 procedures are performed in the Netherlands. Currently, two surgical procedures are performed in clinical practice. Most frequently an endarterectomy is performed using a length incision over the artery, followed by a patch plasty (CEAP), in order to reduce the risk of restenosis. As an alternative the eversion technique (ET) was introduced, in which transversal arteriotomy is performed and the plaque is removed from within. After reconstruction with a patch a >50% restenosis has been described in 6-36% of patients during long-term follow-up. When using the eversion technique this is seen in 1.7-2.5%, while also the risk on adverse events seem to be lower. One of the drivers for atherosclerosis in general is a disturbance of local blood flow. This may lead to turbulence, recirculation and stasis of blood. The subsequent low Wall Shear Stress may lead to the ne formation of plaque that in turn may become instable and cause recurrent ischemic events. Recently, a breakthrough was achieved in the imaging options of flow in the carotid arteries, using Vector Flow Imaging. Using a fully programmable ultrasound machine, over 10,000 frames per second can be captured, in comparison to about 50 in regular ultrasound. This enables the tracking of particles that, after processing will provide the needed flow information. A recent study, comparing flow before and after CEAP has shown that there is significant recirculation after reconstruction. This raises the question whether this would be more optimal after ET, which would support the potential lower incidence of recurrent stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Presence of carotid artery stenosis (≥50%) according to conventional clinically performed imaging (duplex/CT(A)/MR(A)) for which patient underwent uncomplicated CEA with either a patch plasty or the eversion technique
* ≥18 years old;
* Able to provide signed or oral informed consent
* Carotid artery <25mm below skin

Exclusion Criteria:

* Carotid bifurcation with depth of center bulb lumen ≥2.5cm
* Restenosis after carotid revascularisation at side of interest
* Participating in another clinical study, interfering on outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that underwent a CEA, without residual stenosis after surgery, will be included in this study. Patients with ET will be recruited in two collaborating hospitals (ETZ and MST) at the department of Vascular Surgery. Participants to the CAP-VALUE trial (Rijnstate and Radboud) are included, where already ultrasound measurements after CEAP were acquired.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
2D spatio-temporal blood flow velocity profiles | 6-8 weeks after CEA
  2D vector velocity fields derived from the US-based flow images will be used to calculate the spatio-temporal blood flow velocities.

SECONDARY OUTCOMES:
Wall shear stress | 6-8 weeks after CEA
  Multiple blood flow-related parameters will be derived from the spatio-temporal blood flow velocity data. One parameter is wall shear stress.
Vortex identification | 6-8 weeks after CEA
  Multiple blood flow-related parameters will be derived from the spatio-temporal blood flow velocity data. One parameter is vortex identification.
Vector complexity | 6-8 weeks after CEA
  Multiple blood flow-related parameters will be derived from the spatio-temporal blood flow velocity data. One parameter is vector complexity.

CONTACTS AND LOCATIONS:
Overall Officials: Michel M.P.J. Reijnen, MD, PhD, Principal Investigator — Rijnstate Hospital

IPD SHARING:
Plan to Share IPD: Undecided